CLINICAL TRIAL: NCT06066944
Title: Immediate and Prolonged Effects of Thai Foot Massage on Pain, Range of Motion and Somatosensory Reception Among Patients With Type 2 Diabetes Peripheral Neuropathy.
Brief Title: Effect of Thai Foot Massage on Type 2 Diabetes Peripheral Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Azra Khanum, principal investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Foot Massage RCT 001
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Peripheral Diabetic Neuropathy
Keywords: Peripheral neuropathy; Thai Foot Massage; Range of Motion; Ipswich Touch Test (IpTT); Somatosensory Reception
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to the intervention and control group randomly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The experimental group will receive a Thai Foot Massage every alternate day for 30 minutes for 15 days.
  Interventions: Other: Thai Foot Massage
- Group B (No Intervention): Participants in the control group will continue with the standard treatment regimen prescribed by the physician at the diabetic clinic. Baseline data will be collected as conducted for the experimental group. After the completion of the study, if the intervention will prove effective, the Thai foot massage will be applied to the control group.

INTERVENTIONS:
Other: Thai Foot Massage — It is the application of Massage through specific techniques and pressure to the feet and lower legs to promote relaxation, improve circulation, and enhance overall well-being. It is a traditional therapeutic practice originating from Thailand and is often performed by trained practitioners. Thai foot massage is often based on traditional Thai massage techniques. The researcher is duly certified for the administration of Thai Foot Massage.
  Other Names: Control group will continue with the standard care advised by the physician
  Arms: Group A

SUMMARY:
The goal of this clinical trial is to examine the effect of Thai-Foot Massage on type 2 diabetes peripheral neuropathy. The main question is to answer the role of massage in improving peripheral neuropathy. Thai Foot Massage will be administered by the researcher every alternate day for 15 days. Researchers will compare the intervention group with the control group (without intervention) to see the improvement in Somatosensory Reception, Range of Motion, and peripheral neuropathy-induced Pain.

DETAILED DESCRIPTION:
Type 2 diabetes is a chronic metabolic disorder associated with elevated blood sugar levels and various complications, including peripheral neuropathy. This condition damages the nerves controlling sensation, often leading to foot-related issues such as limited range of motion, pain, and Somatosensory Reception deficit. These foot problems pose a significant concern for individuals with diabetes, affecting their overall foot health. Engaging in physical activity programs has been shown to reduce hospitalizations and severe complications in diabetes patients. Foot massage is a specific physical activity aimed at preventing podiatry issues. The study's hypothesis questions whether Thai Foot Massage has immediate and prolonged effects on foot pain, range of motion, and Somatosensory Reception among patients with Type 2 Diabetes Peripheral Neuropathy. This research seeks to determine the impact of Thai Foot Massage on these parameters. Type 2 diabetes and peripheral neuropathy are growing global health concerns and claim a significant social and financial burden. Diabetes Peripheral Neuropathy (DPN) has an impact on quality of life. This study aims to evaluate non-pharmacological interventions to prevent neuropathic complications, including diabetic foot problems and limb amputation. The research design chosen for this study is a Randomized Controlled Trial, recognized for establishing cause-and-effect relationships. The sample will be collected through a non-probability purposive sampling technique and will consist of individuals diagnosed with Type 2 diabetes experiencing peripheral neuropathy symptoms by calculating IpTT score ≤ 4/6. The study will be done at the University of Health Sciences in collaboration with the Diabetic Clinic District Headquarters Shiekhupura. A sample size of 78 participants, with a 5% attrition rate, will be divided equally between intervention and control groups using randomization through a lottery method. Statistical analysis will be performed using SPSS version 27, describing categorical variables through frequency and percentage. The association of qualitative data will be assessed with Chi-square, while an independent t-test and repeated measures of ANOVA will compare the two groups and measure time effects for normal data. In short, this study aims to enhance our understanding of how Thai Foot Massage can impact pain, range of motion, and somatosensory reception in patients with Type 2 diabetes and peripheral neuropathy. The findings may offer valuable insights into non-pharmacological interventions for improving foot health in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age range, 40 to 65, to ensure a consistent demographic.
* Both genders will be part of the study.
* Participants must have a confirmed medical diagnosis of Type 2 Diabetes by the physician and do not have an ulcer or amputation in either foot.
* A score on the Ipswich touch test less than 4/6 will be included.
* Patients must have a level of glycated hemoglobin HbA1C more than 7.
* Individuals receiving treatment for diabetes mellitus, which may include oral hypoglycemic agents, insulin, or both."

Exclusion Criteria:

* Individuals with pre-existing neurological conditions unrelated to diabetes or peripheral neuropathy.
* Participants having severe diabetic complications such as advanced nephropathy, retinopathy or vascular disease will not be included in the study.
* Individuals with foot ulcers, infections, or any medical conditions that prevent them from receiving foot massage safely

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-01-25 (Estimated); Primary Completion 2025-04-25 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Ipswich Touch Test Score (IpTT) | 1 Months
  To measure the somatosensory level, Ipswich Touch Test (IpTT) is a reliable and valid test to assess the sensory deficit in diabetic-related neuropathy patients. The highest score is 6. 6/6 means no neuropathy and 0/6 means worse possible neuropathy.
Measure the Range of Motion | 1 Months
  Range of motion refers to the extent of movement that can be achieved at a specific joint. In this study, the range of motion of the foot and ankle joints will be measured using goniometry, a technique that involves using a universal goniometer to measure the angles of joint movement. ROM will be assessed for the ankle joint, in degrees of dorsiflexion and plantarflexion.
Measure the intensity of neuropathy induced pain | 1 Month
  Pain is defined as "an unpleasant sensory and emotional experience associated with actual or potential tissue damage, reported by patients. In this study pain refers to the unpleasant sensations caused by type 2 diabetes peripheral neuropathy. Pain will be measured through numeric rating pain scale, which ranges from 0 to 10, where "0" represent No Pain and 10 represent worse possible pain. Pain can categorize according to pain score.
  Mild pain: A score of 1 to 3 Moderate Pain: A score of 4 to 6. Severe Pain: A score of 7 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Azra Khanum, 1, Principal Investigator — PG Nursing

IPD SHARING:
Plan to Share IPD: No